CLINICAL TRIAL: NCT06999486
Title: NEW METHODOLOGIES FOR CUSTOMISING SUPPORT FOR FAMILIES OF CHILDREN WITH DIABETES: Validation of a Computerised Adaptive Test for Measuring Caregiver Well-being
Brief Title: Validation of a Computerised Adaptive Test for Measuring Caregiver Well-being
Status: Completed | Type: Observational
Sponsor: Adhera Health, Inc. (Industry)
Collaborators: Hospital Miguel Servet (Other)
Responsible Party: Sponsor
Other Study IDs: RO01
Record Dates: First submitted 2025-05-23; First posted 2025-05-31 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: T1D
Keywords: Type 1 Diabetes; mhealth; caregiver; CAT
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary caregivers of a child with T1D: Caregivers who are the primary caregivers of a child with T1D.
  Interventions: Other: CAT well-being test

INTERVENTIONS:
Other: CAT well-being test — Evaluate the psychometric properties (e.g., reliability, validity) of the Computerized Adaptive Testing (CAT) system for assessing the well-being of caregivers of children with Type 1 Diabetes (T1D).

SUMMARY:
The main objective of this project is to test whether a tool (questionnaire) is suitable for assessing how caregivers of children and adolescents with TD1 feel emotionally and psychologically. To do this, the investigators will use a technological system called 'Computerised Adaptive Testing' (CAT), which adapts the questions according to the answers of each participant. This allows the investigators to obtain a more accurate assessment tailored to each person's particular situation.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers aged ≥18 years who are the primary caregivers of a child with T1D.
* The child should be younger than 18 years with a confirmed diagnosis of T1D.
* Willingness and ability to use a smartphone-based sensing system.
* Willingness to share retrospective continuous glucose monitoring (CGM) data from the child, specifically from the previous 2 months prior to joining the study.

Exclusion Criteria:

* Caregivers with significant cognitive or physical impairments preventing study participation.
* Inability to read or understand the Spanish language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary caregivers of a child with T1D from Hospital Universitario Miguel Servet in Zaragoza.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2025-05-26 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Validity and reliability of the CAT system - Emotional outcome 1 | Day 1 to Day 15 (Week 2)
  These tend to be sensitive to change in short-term and will include distress assessed by the Depression Anxiety and Stress Scale (DASS-21) and the distress thermometer. Minimum Value: 0. Maximum Value: 63. Interpretation: Higher scores indicate worse outcomes (greater levels of depression, anxiety, and stress).
Validity and reliability of the CAT system - Emotional outcome 2 | Day 1 to Day 15 (Week 2)
  These tend to be sensitive to change in short-term and will include perceived self-efficacy assessment by the General Self-Efficacy Scale (GSE). Minimum Value: 10. Maximum Value: 40. Interpretation: Higher scores indicate better outcomes (greater self-efficacy).
Validity and reliability of the CAT system - Emotional outcome 3 | Day 1 to Day 15 (Week 2)
  Mental Health Continuum Short Form (MHC-SF): This is a 14-item scale that consists of 3 items measuring emotional well-being, 6 items measuring psychological well-being, and 5 items measuring social well-being. Minimum value: 14 Maximum value: 84. Interpretation: Higher scores indicate greater well-being in each domain.
Validity and reliability of the CAT system - Mood assessment | Day 1 to day 15 (Week 2)
  Positive and Negative Affect Schedule (PANAS) Unit of Measure: - Positive Affect (PA) score range: 10-50 (higher scores indicate greater positive affect). - Negative Affect (NA) score range: 10-50 (higher scores indicate greater negative affect). Description: PANAS is a self-report questionnaire measuring two dimensions of mood: positive and negative affect.
Validity and reliability of the CAT system - Distress Assessment | Day 1 to Day 15 (Week 2)
  Distress Thermometer Unit of Measure: Score on a 0-10 scale (higher scores indicate higher distress). Description: The Distress Thermometer is a single-item, self-report tool measuring psychological distress on a 0-10 scale.
Validity and reliability of the CAT system - Emotional outcome 4 | Day 1 to Day 15 (Week 2)
  WHO-5 Well-Being Index: Widely validated index to assess mental well-being. It consists of five statements relating to the past two weeks. Responses are rated on a 6-point scale. Minumum value=0, maximum value= 25. Interpretation: Higher scores indicate better well-being. A raw score below 13 may suggest poor well-being and may warrant further evaluation for depression.

SECONDARY OUTCOMES:
Usability and acceptability of the CAT | Day 15 (Week 2)
  Outcome Measure: System Usability Scale (SUS) score. Unit of Measure: SUS score (0-100, higher scores indicate better usability). Description: The System Usability Scale is a 10-item scale based on a 5-point Likert scale assessing perceived usability.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Miguel Servet, Zaragoza, Aragon, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silverstein J, Klingensmith G, Copeland K, Plotnick L, Kaufman F, Laffel L, Deeb L, Grey M, Anderson B, Holzmeister LA, Clark N; American Diabetes Association. Care of children and adolescents with type 1 diabetes: a statement of the American Diabetes Association. Diabetes Care. 2005 Jan;28(1):186-212. doi: 10.2337/diacare.28.1.186. No abstract available. PMID 15616254
- [Background] Katsarou A, Gudbjornsdottir S, Rawshani A, Dabelea D, Bonifacio E, Anderson BJ, Jacobsen LM, Schatz DA, Lernmark A. Type 1 diabetes mellitus. Nat Rev Dis Primers. 2017 Mar 30;3:17016. doi: 10.1038/nrdp.2017.16. PMID 28358037